CLINICAL TRIAL: NCT03142555
Title: Assessing the Corporate Environment in Promoting Tobacco Control and Evaluation of a Smoking Cessation Programme in Workplaces in Hong Kong
Brief Title: Smoking Cessation Programme in Workplaces in Hong Kong (Phase III)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: LST SCPW P3
Record Dates: First submitted 2017-04-24; First posted 2017-05-05 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health talk plus intensive social media intervention (Experimental): Subjects in this group will receive:
  1. General health talk;
  2. Phone follow-up/counselling service (15 - 30 minutes);
  3. Social media (intensive reminders);
  4. Regular personalized what's app interaction ( up to 2 months duration)
  Interventions: Behavioral: Health talk plus intensive social media intervention
- Health talk plus less intensive social media intervention (Placebo Comparator): Subjects in this group will receive:
  1. General health talk;
  2. Phone follow-up/counselling service (15 - 30 mintues);
  3. Social media ( less intensive reminders)
  Interventions: Behavioral: Health talk plus less intensive social media intervention

INTERVENTIONS:
Behavioral: Health talk plus intensive social media intervention — Subjects in this group will receive treatments including a general health education talk about smoking cessation. Subjects will also get involved in the personalized what's app interaction (up to 2 months duration) to receive social support to quit smoking. The intervention outcomes and subjects' smoking status will be followed up regularly via telephone interviews (15 - 30 minutes).
  Arms: Health talk plus intensive social media intervention
Behavioral: Health talk plus less intensive social media intervention — Subjects in this group will receive treatments including a general health education talk about smoking cessation but without the information of active referral to other smoking cessation services. Subjects will receive less intensive reminders via social media. The intervention outcomes and subjects' smoking status will be followed up regularly via telephone interviews (15 - 30 minutes).
  Arms: Health talk plus less intensive social media intervention

SUMMARY:
Smoking causes cardiovascular and respiratory diseases, cancers and diabetes, and it has been a leading risk factor for death globally. Despite the availability of smoking cessation services locally, most smokers do not use such services. Workplace is one of the most convenient platforms to provide smoking cessation services and over 55% of smokers are employed according to the local population-based survey. However, the effectiveness of a smoking cessation programme conducted in workplace is yet to be examined in Hong Kong, and the attitudes and practices of corporations in promoting smoking cessation are not clear. Thus, this study aims to examine the employers'/managerial staff's knowledge, attitudes and practices in promoting smoking cessation in workplace and evaluate the smoking behaviours of participants before and after attending a smoking cessation intervention.

DETAILED DESCRIPTION:
This study will separate into two phases. Phase I is a large scale cross-sectional survey to corporations in Hong Kong to examine the employers' knowledge, attitudes and practices in promoting smoking cessation in the workplace. Phase II is a randomized controlled trial study to evaluate the effectiveness of a smoking cessation intervention to assess the subjects' smoking behaviors, knowledge on smoking and satisfaction of the smoking cessation services. The investigators are interested to know if the intervention package including health education,social media and telephone follow-up would trigger higher quit rate or other changes in smoking behaviors. The investigators will also monitor the smoking status of the subjects regularly through telephone follow-ups, understand the company's practices about smoke-free policy as well as evaluate the outcomes of the intervention.

The primary outcome of the study is to measure participated smokers' self-reported 7-day point prevalence quit rate at 26 weeks follow-ups. The secondary outcomes include participated smokers' (i) self-reported reduction rate at 52 weeks follow-ups; (ii) self-reported quit attempt at 26 and 52 weeks follow-ups; (iii) self-reported reduction rate at 26 and 52 weeks follow-ups; (iv) Engagement in social media intervention.

Data of the above outcomes will be collected through telephone interviews (follow-ups) by the investigators. Descriptive statistics will be used to measure the (1) basic info of the participants, including the total number of employees and smoking employees; (2) knowledge on smoking of employers/managerial staff; (3) attitudes on smoking cessation of employers/managerial staff; (4) practices of the corporations with respect to smoking cessation. Logistic regression, linear regression and spearman correlation coefficient will be used to examine the relationships between corporates' policy in smoking cessation and the knowledge and attitudes of employers/ managerial staff. Chi square and t-test will also be used to compare the quit rates between groups and logistic regression will be used to predict quitting. Data will be entered and analyzed using IBM SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Cantonese speaker
* Smoke at least one cigarette per day in the past 30 days
* Stay in Hong Kong during the intervention and follow-up periods (12 months)

Exclusion Criteria:

* Smokers who are psychologically or physically unable to communicate
* Currently following other smoking cessation programme(s)
* Smokers with diagnosed psychiatric illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 679 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 26 weeks
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence quit rate | 52 weeks
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Self-reported reduction rate | 26 and 52 weeks
  Smokers' who reduced tobacco use (in term of daily cigarette consumption) in the follow-up when comparing with the baseline
Self-reported quit attempt rate | 26 and 52 weeks
  Smokers' who refrained from smoking for 24 hours in the 7 days preceding the follow-up
Engagement in social media intervention | 26 weeks
  Self-reported engagement in social media intervention in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Study Director — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weng X, Lau OS, Ng CH, Li WHC, Lam TH, Wang MP. Effect of a workplace mobile phone-based instant messaging intervention on smoking cessation: a cluster-randomized controlled trial. Addiction. 2022 Jun;117(6):1758-1767. doi: 10.1111/add.15804. Epub 2022 Feb 6. PMID 35037319